CLINICAL TRIAL: NCT00088959
Title: Phase I Study of Erlotinib and Celecoxib in Former Smokers With Advanced Non-Small Cell Lung Cancer
Brief Title: Celecoxib and Erlotinib in Treating Former Smokers With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00886; 4939-04-6R2; DUMC-4939-03-6R0; VAMC-DURHAM-00813; DUMC-GCRC-911; CDR0000377689; DUMC-4939-04-6R2; U01CA096123 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (erlotinib hydrochloride, celecoxib) (Experimental): Patients receive oral erlotinib hydrochloride once daily and oral celecoxib twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: celecoxib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: celecoxib — Given orally
  Other Names: Celebrex; SC-58635
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of celecoxib when given together with erlotinib in treating former smokers with stage IIIB, stage IV, recurrent, or progressive non-small cell lung cancer. Celecoxib and erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the clinical toxicity and tolerability of erlotinib combined with celecoxib in patients with advanced non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To estimate the tumor response rate of erlotinib combined with celecoxib in patients with advanced NSCLC.

II. To estimate the dose of celecoxib that results in maximal induction of apoptosis, maximal inhibition of prostaglandin E2 (PGE2) in bronchoalveolar (BAL) fluid, and maximal inhibition of bronchial cell proliferation when combined with erlotinib.

III. To estimate the effect of erlotinib and the combination of erlotinib and celecoxib on bronchial expression of COX-2.

IV. To estimate the effect of erlotinib and the combination of erlotinib (and celecoxib on autophosphorylation of epidermal growth factor receptor (EGFR) in skin and endobronchial biopsies.

V. To estimate the degree of correlation of autophosphorylation of EGFR in skin and endobronchial samples.

TERTIARY OBJECTIVES:

I. To estimate the effect of the combination of erlotinib and COX-2 inhibitor (celecoxib) on the frequency of fractional allelic loss (FAL) in endobronchial biopsies, metaplasia and dysplasia in endobronchial biopsies, and endobronchial proliferation.

OUTLINE: This is an open-label, dose-escalation study of celecoxib.

Patients receive oral erlotinib hydrochloride once daily and oral celecoxib twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of celecoxib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 6 additional patients are treated at the MTD.

Patients are followed at 4 weeks.

ELIGIBILITY:
Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) meeting 1 of the following stage criteria: Stage IIIB with pleural effusion; Stage IV disease; recurrent or progressive disease after prior surgery, radiotherapy, and/or chemotherapy
* If the sole prior treatment was in the adjuvant or neoadjuvant setting, tumor progression or recurrence must have occurred within 6 months after completion of prior treatment
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 g/dL
* Hemostasis normal
* Creatinine =< 2.0 mg/dL
* No significant cardiovascular disease
* No New York Heart Association class III or IV cardiac disease
* No uncontrolled dysrhythmia
* No unstable angina
* No myocardial infarction within the past 6 months
* FEV1 >= 1.0 liter OR 40% of predicted within the past 3 months
* Oxygen saturation >= 90% on room air
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study treatment
* Willing to undergo bronchoscopy
* No allergy to sulfonamides or hypersensitivity reaction to celecoxib
* No other medical or psychological condition (e.g., acute psychosis) that would preclude study participation
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin)
* At least 4 weeks since prior radiotherapy
* Prior complete resection allowed provided there is histologic and cytologic documentation of disease recurrence
* More than 3 months since prior chemopreventative agents (e.g., oltipraz, retinoids, or N-acetylcysteine [NAC])
* No prior erlotinib hydrochloride
* No other prior EGFR antagonists
* No concurrent medication known to interact with erlotinib hydrochloride or celecoxib, including the following: Fluconazole, Lithium, Furosemide, Angiotensin-converting enzyme inhibitors, Phenytoin, Carbamazepine, Rifampin, Barbiturates, Hypericum perforatum (St. John's wort)
* No concurrent non-steroidal anti-inflammatory drugs
* Concurrent aspirin of up to an average dose of 325 mg/day allowed
* No aspirin treatment for 7 days prior to any bronchoscopic or skin biopsy
* No other concurrent EGFR inhibitors or cyclo-oxygenase-2 (COX-2) inhibitors
* Meets 1 of the following criteria: 1) Advanced NSCLC with at least stable disease after >= 4 courses of platinum-containing chemotherapy 2) Relapsed or refractory disease after treatment with >= 1 prior platinum-containing chemotherapy program, including adjuvant or neoadjuvant therapy for NSCLC
* No untreated brain metastases
* ECOG 0-1
* Former smoker, as indicated by the following: 1) At least a 30 pack-year smoking history 2) Smoking duration at least 10 years 3) At least 12 months of self-reported smoking cessation 4) Negative urine cotinine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-12; Primary Completion 2009-01 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Clinical tolerable dose of celecoxib as measured by NCI CTCAE v3.0 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kelley, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States